CLINICAL TRIAL: NCT00319501
Title: A Phase 3, Randomized, Double-blind, Parallel, Placebo-controlled, Multicenter Study, With Optional Open-label Continuation, Of The Efficacy And Safety Of Vanquix(tm) Auto-injector (Diazepam Injection) For The Management Of Selected, Refractory, Patients With Epilepsy Who Require Intermittent Medical Intervention To Control Episodes Of Acute Repetitive Seizures
Brief Title: Efficacy and Safety of Diazepam in the Management of Refractory Epilepsy in Selected Patients Who Require Intermittent Medical Intervention for Acute Repetitive Seizures.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K826-05-3001; B4511001 (Other: Alias Study Number); NCT01079156 (obsolete NCT alias)
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Results first posted 2016-08-16 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-07

CONDITIONS: Seizures; Epilepsies, Partial; Epilepsy, Complex Partial; Epilepsy, Generalized; Epilepsy
Keywords: Acute Repetitive Seizures; ARS; Diazepam; Cluster Seizures
MeSH Terms: conditions — Seizures; Epilepsies, Partial; Epilepsy, Complex Partial; Epilepsy, Generalized; Epilepsy | interventions — Diazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): During the Double-blind Period, participants received a single, age- and weight-appropriate dose of placebo solution as a deep intramuscular injection in the mid to outer thigh. Drug was administered by a caregiver using a spring-driven, pressure-activated, prefilled autoinjector at the onset of an episode of acute repetitive seizures (ARS).
  Interventions: Drug: Placebo
- Diazepam (Experimental): During the Double-blind Period, participants received a single, age- and weight-appropriate dose of diazepam solution, ranging from 0.2 to 0.5 mg/kg, as a deep intramuscular injection in the mid to outer thigh. Additional doses were permissible during the Open-label Period. Drug was administered by a caregiver using a spring-driven, pressure-activated, prefilled autoinjector at the onset of an episode of ARS.
  Interventions: Drug: Vanquix Auto-Injector (Diazepam Injection)

INTERVENTIONS:
Drug: Placebo — Intramuscular autoinjector; administered at onset of an episode
  Arms: Placebo
Drug: Vanquix Auto-Injector (Diazepam Injection) — Intramuscular autoinjector: 5, 10, 15, or 20 mg (based on participant's age and weight); administered at the onset of an episode
  Arms: Diazepam

SUMMARY:
To evaluate the efficacy and safety of diazepam in the management of refractory epilepsy in selected patients who require intermittent medical intervention for the control of episodes of acute repetitive seizures. In addition, to assess the support provided by caregivers who are not themselves or not under the direct supervision of health care professionals at the time of administration.

ELIGIBILITY:
Key Inclusion Criteria

For Patient:

* Older than 2 years of age and between 6 and 136 kg body weight
* Recipient of clinical diagnosis of epilepsy, taking a stable antiepileptic drug regimen for at least 2 weeks, and requiring intermittent medical intervention to control episodes of acute repetitive seizures (ARS)
* Experienced at least 2 episodes of ARS in previous year, one of which occurred in previous 6 months
* Has episodes of ARS that include complex partial or generalized seizures
* Has a responsible caregiver available to participate
* Is not pregnant or lactating and is practicing an acceptable method of birth control.

For Caregiver:

* Age of 18 years or older and has demonstrated responsibility as a caregiver through training to:

  * Recognize an episode of repetitive seizures for which the injection was intended,
  * Administer study drug
  * Count and record seizures and respiratory rate in the patient diary,
  * Monitor the patient and record observations in the patient diary for 12 hours following study drug treatment
  * Recognize the need for immediate medical attention.

Key Exclusion Criteria

For Patient:

* Petit mal status or petit mal variant status
* History of ARS consistently progressing to status epilepticus
* History of failure to respond to benzodiazepine treatment
* Hypersensitivity to diazepam
* Acute narrow angle glaucoma
* Alcohol and/or other substance abuse
* Has taken another investigational drug in previous 30 days
* Acute or progressive neurologic or severe psychiatric disease or severe mental abnormality.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2006-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (85):
- United States (85):
  - Neurology Clinic, PC, Northport, Alabama
  - Clinical Trials, Inc, Little Rock, Arkansas
  - Stein Life Child Neurology Medical Specialists Inc., Irvine, California
  - Collaborative NeuroScience Network, LLC, Long Beach, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Brain and Spine Surgeons of Orange County, Newport Beach, California
  - Drug Shipment, Sacramento, California
  - Sacramento Comprehensive Epilepsy Program, Sacramento, California
  - Sutter Cancer Center Specialty Clinic, Sacramento, California
  - Sutter Institute for Medical Research, Sacramento, California
  - Northern California Cardiology, Sacramento, California
  - Bradenton Research Center, Inc., Bradenton, Florida
  - Morton Plant Hospital Epilepsy Clinic, Clearwater, Florida
  - Morton Plant Hospital Pharmacy, Clearwater, Florida
  - Child Neurology Center of NorthWest Florida, Gulf Breeze, Florida
  - NorthWest Florida Clinical Research Group, LLC, Gulf Breeze, Florida
  - Emery Neuroscience Center, Lighthouse PT, Florida
  - Pediatric Neurology and Epilepsy Center, Loxahatchee Groves, Florida
  - Miami Children's Hospital, Miami, Florida
  - EKG only, Orlando, Florida
  - Pediatric Neurology, PA, Orlando, Florida
  - AMO Corp, Tallahassee, Florida
  - Tallahassee Neurological Clinic, Tallahassee, Florida
  - Pediatric Epilepsy & Neurology Specialists, Tampa, Florida
  - Willsey Research Inc, Tampa, Florida
  - Child Neurology Associates, PC, Atlanta, Georgia
  - Savannah Neurology, PC, Savannah, Georgia
  - Consultants in Epilepsy and Neurology, PLLC, Boise, Idaho
  - Comer Children's Hospital, Chicago, Illinois
  - University of Chicago Hospital Pharmacy, Chicago, Illinois
  - University of Chicago Medical Center (UCMC) Center for Advanced Medicine (CAM), Chicago, Illinois
  - University of Chicago Medical Center (UCMC), Chicago, Illinois
  - University Neurologists PSC Pediatric Division, Louisville, Kentucky
  - University of Louisville Ambulatory Care Building Clinic, Louisville, Kentucky
  - University of Louisville Clinical Trials Unit, Louisville, Kentucky
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - Neurology Clinic of St Cloud, Saint Cloud, Minnesota
  - The Comprehensive Epilepsy Care Center For Children and Adults, Chesterfield, Missouri
  - MRI Location, Kansas City, Missouri
  - St Luke's Hospital Neurological Consultants, Kansas City, Missouri
  - St Luke's Hospital, Kansas City, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Clinical Research Center of New Jersey, Gibbsboro, New Jersey
  - University of Medicine and Dentistry of New Jersey Robert Wood Johnson Medical Group, New Brunswick, New Jersey
  - University of Medicine and Dentistry of New Jersey-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Elmwood Clinic, Buffalo, New York
  - Millard Fillmore Gates Hospital/Comprehensive Epilepsy Center, Buffalo, New York
  - Women and Children's Hospital of Buffalo, Buffalo, New York
  - NYU Medical Center, Comprehensive Epilepsy Center, New York, New York
  - Strong Memorial Hospital, Rochester, New York
  - University of Rochester, Strong Epilepsy Center, Rochester, New York
  - Cone Health Child Neurology, Greensboro, North Carolina
  - Guilford Neurologic Associates, Greensboro, North Carolina
  - Raleigh Neurology Associates, PA, Raleigh, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Cleveland Clinic Health Systems, Cleveland, Ohio
  - Ohio State University Neurology Clinic, Columbus, Ohio
  - Ohio State University University Hospital, Columbus, Ohio
  - Ohio State University, Columbus, Ohio
  - North Pacific Epilepsy Research/The Northrup Center, Portland, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Wellspan Neurosciences, York, Pennsylvania
  - Apple Hill Medical Center (EKG & Lab Draw), York, Pennsylvania
  - Medical University of South Carolina Hospitals and Clinics, Charleston, South Carolina
  - Medical University of South Carolina/Department of Pharmacy Service, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - The Neurology and Pain Clinic, Orangeburg, South Carolina
  - Mid-South Physicians Group, PLLC, Germantown, Tennessee
  - University of Tennessee Lebonheur Pediatric Specialists Inc., Memphis, Tennessee
  - Access Clinical Trial, Inc., Nashville, Tennessee
  - CMC - Physician's Park, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Vanderbilt Epilepsy Clinic, Nashville, Tennessee
  - Vanderbilt University Hospital Pharmacy, Nashville, Tennessee
  - Neurological Clinic of Texas, PA, Dallas, Texas
  - Cook Children's Medical Center Office of Grants and Research, Fort Worth, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Cook Children's Physcian Network, Fort Worth, Texas
  - Alamo City Clinical Research, LLC, San Antonio, Texas
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - Virginia Commonwealth University Division of Child Neurology, Richmond, Virginia
  - Virginia Commonwealth University Ambulatory Care Center/Department of Neurology, Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington
  - University of Washington Regional Epilepsy Center, Harborview Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Abou-Khalil B, Wheless J, Rogin J, Wolter KD, Pixton GC, Shukla RB, Sherman NA, Sommerville K, Goli V, Roland CL. A double-blind, randomized, placebo-controlled trial of a diazepam auto-injector administered by caregivers to patients with epilepsy who require intermittent intervention for acute repetitive seizures. Epilepsia. 2013 Nov;54(11):1968-76. doi: 10.1111/epi.12373. Epub 2013 Sep 20. PMID 24111974
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=K826-05-3001&StudyName=Efficacy%20and%20safety%20of%20Vanquix%20for%20the%20management%20of%20selected%2C%20refractory%2C%20patients%20with%20epilepsy%20who%20require%20intermittent%20caregiver

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 234 participants randomized, 71 (29 placebo, 42 diazepam) did not receive/attempt to receive treatment. Discontinuation prior to treatment due to: 3,0 protocol violations; 6,5 sponsor's request; 4,8 Principal Investigator request; 5,11 other; 0,2 lost to follow-up, and 9,10 withdrawn consent.
Groups:
- Diazepam: During the Double-blind Period, participants received a single, age- and weight-appropriate dose of diazepam solution, ranging from 0.2 to 0.5 mg/kg, administered by caregivers untrained as and unsupervised by healthcare professionals. Drug was delivered by a spring-driven, pressure-activated, prefilled autoinjector at the onset of an episode of acute repetitive seizures (ARS). Additional doses were permissible as needed during the Open-label and Open-label Extension Periods.
- Placebo: During the Double-blind Period, participants received a single, age- and weight-appropriate dose of placebo solution as a deep intramuscular injection in the mid to outer thigh. Drug was administered by a caregiver using a spring-driven, pressure-activated, prefilled autoinjector at the onset of an episode of ARS.
Period: Double-blind Period
Arm/Group | Diazepam | Placebo
Started | 124 (Randomized participants) | 110 (Randomized participants)
Received Treatment | 82 | 81
Completed | 81 | 78
Not Completed | 43 | 32
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Sponsor Request | 1 | 0
Not completed — Did not receive treatment | 42 | 29
Period: Open-label Period
Arm/Group | Diazepam | Placebo
Started | 161 (Participants who continued to meet eligibility requirements) | 0
Received Treatment | 128 | 0
Completed | 45 (Competed=continuing treatment) | 0
Not Completed | 116 | 0
Not completed — Adverse Event | 5 | 0
Not completed — Protocol Violation | 6 | 0
Not completed — Withdrawal by Subject | 38 | 0
Not completed — Principal Investigator decision | 6 | 0
Not completed — Sponsor request | 12 | 0
Not completed — Lost to Follow-up | 5 | 0
Not completed — Did not receive treatment | 33 | 0
Not completed — Other | 11 | 0
Period: Open-label Extension Period
Arm/Group | Diazepam | Placebo
Started | 51 (Eligible participants who chose to continue treatment) | 0
Received Treatment | 33 | 0
Completed | 0 | 0
Not Completed | 51 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Did not receive treatment | 18 | 0
Not completed — Other | 1 | 0
Not completed — Principal investigator decision | 2 | 0
Not completed — Sponsor request | 26 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: Participants who were randomized to receive treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Diazepam | Placebo | Total
Number analyzed (Participants) | 124 | 110 | 234
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.8 (15.98) | 21.3 (12.92) | 22.1 (14.61)
Age, Customized [Number; unit: participants]
  2 to 5 years | 12 | 6 | 18
  6 to 11 years | 18 | 14 | 32
  12 years and older | 94 | 90 | 184
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 54 | 116
  Male | 62 | 56 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 9 | 24
  Not Hispanic or Latino | 109 | 101 | 210
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White/Caucasian | 104 | 89 | 193
  Black/African American | 13 | 17 | 30
  Asian | 2 | 2 | 4
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0
  Other | 5 | 2 | 7
  Missing | 0 | 0 | 0
Place of Residence [Number; unit: Participants]
  Home | 123 | 107 | 230
  Foster home | 0 | 1 | 1
  Group home | 1 | 1 | 2
  Residential facility | 0 | 1 | 1
  Other | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: Centimeters] | 154.2 (25.08) | 154.5 (22.61) | 154.4 (23.91)
Weight [Mean (Standard Deviation); unit: Kilograms] | 61.0 (29.15) | 58.9 (28.47) | 60.0 (28.79)

OUTCOME MEASURES:

1. Primary Outcome: Time to Next Seizure or Rescue Medication During the Double-blind Period (Kaplan-Meier 50th Percentile)
Description: An event was defined as an episode of or required rescue medication for an episode of acute repetitive seizures (ARS) within 15 minutes to 12 hours following study drug administration. Patients without an ARS event were censored at 12 hours. Diaries were provided; if no diary was returned, or the diary did not provide answers to questions about seizures and rescue during the 12-hour follow-up period, the patient was considered censored as of 15 minutes past the treatment time, unless another contact was documented. If seizure control following study drug administration was inadequate, diazepam rectal gel was provided as a rescue medication, given only in the first 4 hours after study drug administration and only if the caregiver was directed to do so by the Investigator or designee at the time of the ARS episode. Patients and their caregivers were trained to recognize the onset of an episode of ARS and when and how to administer study drug.
Time Frame: From 15 minutes to 12 hours after study drug administration for an episode of ARS during the Double-blind Period
Population: All randomized participants for whom an attempt (successful or not) was made to administer study drug for an ARS event during the Double-blind Period.
Measure: Median (95% Confidence Interval); unit: Hours
Groups:
- Diazepam: Participants received a single, age- and weight-appropriate dose of diazepam solution, ranging from 0.2 to 0.5 mg/kg, administered by caregivers untrained as and unsupervised by healthcare professionals. Drug was delivered by a spring-driven, pressure-activated, prefilled autoinjector at the onset of an episode of acute repetitive seizures (ARS).
Arm/Group | Diazepam | Placebo
Number analyzed (Participants) | 82 | 81
Hours | 5.92 [2.28 to NA] — NA=not available. Not estimable due to the low number of events in the arm | NA [NA to NA] — NA=not available. Not estimable due to the low number of events in the arm
Statistical Analysis 1: Comparison: Diazepam; Null hypothesis; Test type: Superiority or Other; p = 0.012, Cox Proportional Hazard — p-value is adjusted. All statistical tests were 2-sided and employed a level of significance of alpha=0.05; Hazard Ratio (HR) = 0.55, 95% CI 2-sided [0.34 to 0.88] — Age adjusted

2. Primary Outcome: Percentage of Participants With an Event (Next Seizure or Rescue Medication) During the Open-label Period
Description: as for outcome 1
Time Frame: From 15 minutes to 12 hours after study drug administration for an episode of ARS during the Double-blind Period
Population: All randomized participants for whom an attempt (successful or not) was made to administer study drug for an ARS event during the Open-label Period.
Measure: Number; unit: Percentage of participants
Arm/Group | Diazepam
Number analyzed (Participants) | 129
Percentage of participants | 22.4 [NA to NA]

3. Secondary Outcome: Number of Participants Requiring Rescue Medication During the Double-blind Period
Description: If seizure control following study drug administration was inadequate, diazepam rectal gel was provided as a rescue medication, given only in the first 4 hours after study drug administration and only if the caregiver was directed to do so by the Investigator or designee at the time of the acute repetitive seizure (ARS) episode. Each patient's specific criteria for seizure and an episode of ARS were determined by the Investigator. Patients and their caregivers were trained to use these criteria to recognize the onset of an episode of ARS and when and how to administer study drug. An episode of ARS was defined as an episode of multiple complex, partial, or generalized seizures occurring over a brief period (minutes to 12 hours) with the patient regaining consciousness between seizures, which were readily recognizable by the patient or a trained caregiver. ARS includes seizures sometimes referred to as serial, cluster, crescendo, or stuttering prolonged.
Time Frame: From 15 minutes to 12 hours following study drug administration for an episode of ARS during the Double-blind Period
Population: All randomized participants for whom an attempt (successful or not) was made to administer study drug for an ARS during the Double-blind Period.
Measure: Number; unit: Participants
Groups:
- Diazepam: Participants received an age- and weight-appropriate dose of diazepam solution, ranging from 0.2 to 0.5 mg/kg, administered by caregivers untrained as and unsupervised by healthcare professionals. Drug was delivered by a spring-driven, pressure-activated, prefilled autoinjector at the onset of an episode of acute repetitive seizures (ARS).
Arm/Group | Diazepam | Placebo
Number analyzed (Participants) | 82 | 81
Participants | 14 | 24
Statistical Analysis 1: Comparison: Diazepam; Test type: Superiority or Other; p = 0.066, Fisher Exact — p-value is unadjusted. All statistical tests were 2-sided and employed a level of significance of alpha=0.05

4. Secondary Outcome: Number of Participants Requiring Emergency Department Visits During the Double-blind Period
Description: Any use of emergency treatment (such as an emergency room visit) was recorded in the patient's diary, along with the date, time, and reason for the emergency treatment. Emergency department visits required some type of rescue action taken, other than the visit itself. An episode of acute repetitive seizures (ARS) was defined as an episode of multiple complex, partial, or generalized seizures occurring over a brief period (minutes to 12 hours) with the patient regaining consciousness between seizures, which were readily recognizable by the patient or a trained caregiver. ARS includes seizures sometimes referred to as serial, cluster, crescendo, or stuttering prolonged.
Time Frame: From 15 minutes to 12 hours following study drug administration for onset of an episode of ARS during the Double-blind Period
Population: All randomized participants for whom an attempt (successful or not) was made to administer study drug for an episode of ARS during the Double-blind Period.
Measure: Number; unit: Participants
Arm/Group | Diazepam | Placebo
Number analyzed (Participants) | 82 | 81
Participants | 2 | 4
Statistical Analysis 1: Comparison: Diazepam; Test type: Superiority or Other; p = 0.443, Fisher Exact

5. Secondary Outcome: Number of Participants Requiring Rescue Medical Care Other Than Rescue Medication or Emergency Department Visits During the Double-blind Period
Description: Other rescue medical care consisted of care other than rescue medication or emergency department visits. Each patient's specific criteria for seizure and an episode of acute repetitive seizure (ARS) were determined by the Investigator. Patients and their caregivers were trained to use these criteria to recognize the onset of an episode of ARS and when and how to administer study drug. An episode of ARS was defined as an episode of multiple complex, partial, or generalized seizures occurring over a brief period (minutes to 12 hours) with the patient regaining consciousness between seizures, which were readily recognizable by the patient or a trained caregiver. ARS includes seizures sometimes referred to as serial, cluster, crescendo, or stuttering prolonged.
Time Frame: From 15 minutes to 12 hours following study drug administration for an episode of ARS during the Double-blind Period
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Diazepam | Placebo
Number analyzed (Participants) | 82 | 81
Participants | 0 | 2
Statistical Analysis 1: Comparison: Diazepam; Test type: Superiority or Other; p = 0.245, Fisher Exact — p-value is unadjusted. All statistical tests were 2-sided and employed a level of significance of alpha=0.05

6. Secondary Outcome: Mean Score on Caregiver Global Treatment Assessment During the Double-blind Period
Description: Caregiver global evaluation is based on seizure frequency, severity, and overall outcome compared with previous episodes and is rated on a 10-cm visual analogue scale, where 0=much worse and 10=much better. A higher score indicates greater improvement. An episode of acute repetitive seizures (ARS) is defined as an episode of multiple complex, partial, or generalized seizures occurring over a brief period (minutes to 12 hours) with the patient regaining consciousness between seizures, which were readily recognizable by the patient or a trained caregiver. ARS includes seizures sometimes referred to as serial, cluster, crescendo, or stuttering prolonged.
Time Frame: Assessments completed at the end of each treated episode of ARS in the Double-blind Period
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Diazepam | Placebo
Number analyzed (Participants) | 79 | 78
Units on a scale | 6.2 (2.79) | 5.5 (2.86)
Statistical Analysis 1: Comparison: Diazepam; Test type: Superiority or Other; p = 0.086, ANOVA — p-Value is unadjusted. All statistical tests were 2-sided and employed a level of significance of alpha = 0.05; ANOVA=analysis of variance; Difference in least square means = 0.75, 95% CI 2-sided [-0.11 to 1.61] — Model included treatment and age category

7. Secondary Outcome: Mean Score on Physician Global Treatment Assessment During the Double-blind Period
Description: Physician global evaluation is based on seizure frequency, severity, and overall outcome compared with previous episodes. The physician global evaluation is rated on a 10-cm visual analogue scale, where 0=much worse and 10=much better. A higher score indicates greater improvement. An episode of acute repetitive seizures (ARS) was defined as an episode of multiple complex, partial, or generalized seizures occurring over a brief period (minutes to 12 hours) with the patient regaining consciousness between seizures, which were readily recognizable by the patient or a trained caregiver. ARS includes seizures sometimes referred to as serial, cluster, crescendo, or stuttering prolonged.
Time Frame: At Visit 2 and subsequent visits in the Double-blind Period
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Diazepam | Placebo
Number analyzed (Participants) | 81 | 78
Units on a scale | 6.3 (2.45) | 5.5 (2.69)
Statistical Analysis 1: Comparison: Diazepam; Test type: Superiority or Other; p = 0.045, ANOVA — p-value is unadjusted. All statistical tests were 2-sided and employed a level of significance of alpha=0.05; Difference in least square means = 0.79, 95% CI 2-sided [0.02 to 1.56] — Model included treatment and age category

8. Secondary Outcome: Number of Participants Requiring Rescue Medication During the Open-label Period
Description: Each patient's specific criteria for seizure and an episode of acute repetitive seizure (ARS) were determined by the Investigator. Patients and their caregivers were trained to use these criteria to recognize the onset of an episode of ARS and when and how to administer study drug. If seizure control following study drug administration was inadequate, diazepam rectal gel was provided as a rescue medication, given only in the first 4 hours after study drug administration and only if the caregiver was directed to do so by the Investigator or designee at the time of the ARS episode.
Time Frame: From 15 minutes to 12 hours after study drug administration during the Open-label Period
Population: All randomized participants in whom an attempt (successful or not) was made to administer study drug for an ARS episode during the Open-label Period of the study.
Measure: Number; unit: Participants
Groups:
- Diazepam: Participants received an age- and weight-appropriate dose of diazepam solution, ranging from 0.2 to 0.5 mg/kg, administered by caregivers untrained as and unsupervised by healthcare professionals. Drug was delivered by a spring-driven, pressure-activated, prefilled autoinjector at the onset of an episode of acute repetitive seizures (ARS). Additional doses were permissible during this period.
Arm/Group | Diazepam
Number analyzed (Participants) | 129
Participants | 39

9. Secondary Outcome: Number of Participants Requiring Emergency Department Visits During the Open-label Period
Description: Any use of emergency treatment (such as an emergency room visit) was recorded in the patient's diary, along with the date, time, and reason for the emergency treatment. Emergency department visits required some type of rescue action taken, other than the visit itself.
Time Frame: From 15 minutes to 12 hours after study drug administration for onset of an episode of ARS during the Open-label Period
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Diazepam
Number analyzed (Participants) | 129
Participants | 13

10. Secondary Outcome: Number of Participants Requiring Rescue Medical Care Other Than Medication or Emergency Department Visits During the Open-label Period
Description: Other rescue medical care consisted of care other than rescue medication or emergency department visits. Each patient's specific criteria for seizure and an episode of acute repetitive seizure (ARS) were determined by the Investigator. Patients and their caregivers were trained to use these criteria to recognize the onset of an episode of ARS and when and how to administer study drug.
Time Frame: From 15 minutes to 12 hours after study drug administration for onset of an episode of ARS during the Open-label Period
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Diazepam
Number analyzed (Participants) | 129
Participants | 5

11. Secondary Outcome: Mean Score on Caregiver Global Treatment Assessment During the Open-label Period
Description: as for outcome 6
Time Frame: Assessments completed at the end of each treated episode of ARS in the Open-label Period
Population: All randomized participants for whom an attempt (successful or not) was made to administer study drug for an ARS event during the Open-label Period and who were available for participation.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Diazepam
Number analyzed (Participants) | 124
Units on a scale | 6.78 (1.896)

12. Secondary Outcome: Mean Score on Physician Global Treatment Assessment During the Open-label Period
Description: Physician global evaluation is based on seizure frequency, severity, and overall outcome compared with previous episodes and is rated on a 10-cm visual analogue scale, where 0=much worse and 10=much better. A higher score indicates greater improvement. An episode of acute repetitive seizures (ARS) is defined as an episode of multiple complex, partial, or generalized seizures occurring over a brief period (minutes to 12 hours) with the patient regaining consciousness between seizures, which were readily recognizable by the patient or a trained caregiver. ARS includes seizures sometimes referred to as serial, cluster, crescendo, or stuttering prolonged.
Time Frame: From Visit 2 and subsequent visits in the Open-label Period to discharge or study termination
Population: All randomized participants for whom an attempt (successful or not) was made to administer study drug for an ARS event during the Open-label Period and who were available for evaluation.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Diazepam
Number analyzed (Participants) | 124
Units on a scale | 6.87 (1.645)

ADVERSE EVENTS:
Description: An adverse event is any untoward unfavorable unintended sign, symptom, or disease temporally associated with the use of drug, whether or not considered related to that drug. A serious adverse event is any untoward medical occurrence that results in death or disability/incapacity; is life-threatening; or requires or prolongs hospitalization.
Groups:
- Diazepam (Double-blind Period): Participants received a single, age- and weight-appropriate dose of diazepam solution, ranging from 0.2 to 0.5 mg/kg, administered by caregivers untrained as and unsupervised by healthcare professionals. Drug was delivered by a spring-driven, pressure-activated, prefilled autoinjector at the onset of an episode of ARS.
- Diazepam (Open-label Period): Participants received an age- and weight-appropriate dose of placebo solution administered using a spring-driven, pressure-activated, prefilled autoinjector. Additional doses were permissible as needed.
- Diazepam (Open-label Extension): Participants continued to receive diazepam in an age- and weight-appropriate dose of administered using a spring-driven, pressure-activated, prefilled autoinjector. Additional doses were permissible as needed at the onset of an ARS episode. Participants were to continue until drug became marketed.
- Placebo (Double-blind Period): Participants received a single dose of diazepam-matching solution as a deep intramuscular injection in the mid to outer thigh. Drug was administered by a caregiver using a spring-driven, pressure-activated, prefilled autoinjector at the onset of an episode of ARS.
Arm/Group | Diazepam (Double-blind Period) | Diazepam (Open-label Period) | Diazepam (Open-label Extension) | Placebo (Double-blind Period)
Serious Adverse Events (participants affected / at risk) | 2/81 | 20/128 | 11/33 | 3/79
Other Adverse Events (participants affected / at risk) | 33/81 | 43/128 | 20/33 | 32/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diazepam (Double-blind Period) (N=81) | Diazepam (Open-label Period) (N=128) | Diazepam (Open-label Extension) (N=33) | Placebo (Double-blind Period) (N=79)
GAIT DISTURBANCES (General disorders) | 1 | 0 | 1 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 | 0 | 0 | 1
EPILEPSY (Nervous system disorders) | 0 | 10 | 5 | 1
HEADACHE (Nervous system disorders) | 0 | 1 | 0 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1 | 0 | 0
STATUS EPILEPTICUS (Nervous system disorders) | 0 | 1 | 1 | 0
POSTICTAL STATE (Nervous system disorders) | 0 | 0 | 1 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
GASTROINTESTINAL STOMA COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
HEAT STROKE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
JAW FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
CORNEAL ABRASION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
AFFECTIVE DISORDER (Psychiatric disorders) | 0 | 1 | 0 | 0
ANXIETY DISORDER (Psychiatric disorders) | 0 | 1 | 0 | 0
DEPRESSION (Psychiatric disorders) | 0 | 1 | 1 | 0
HALLUCINATION, AUDITORY (Psychiatric disorders) | 0 | 1 | 0 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 1 | 0 | 0
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 | 1 | 0 | 0
SUICIDAL IDEATION (Psychiatric disorders) | 0 | 1 | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
PYREXIA (General disorders) | 0 | 1 | 1 | 0
SEPSIS (Infections and infestations) | 0 | 1 | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 0 | 1 | 0 | 0
APPENDICITIS PERFORATED (Infections and infestations) | 0 | 0 | 1 | 0
CELLULITIS (Infections and infestations) | 0 | 0 | 1 | 0
CELLULITIS ORBITAL (Infections and infestations) | 0 | 0 | 1 | 0
HORDEOLUM (Infections and infestations) | 0 | 0 | 1 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
ANGINA PECTORIS (Cardiac disorders) | 0 | 0 | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 0 | 0 | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 1 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 1 | 0
NEPHROTIC SYNDROME (Renal and urinary disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Diazepam (Double-blind Period) (N=81) | Diazepam (Open-label Period) (N=128) | Diazepam (Open-label Extension) (N=33) | Placebo (Double-blind Period) (N=79)
INJECTION SITE PAIN (General disorders) | 14 | 15 | 2 | 11
INJECTION SITE HEMORRHAGE (General disorders) | 4 | 12 | 0 | 5
INJECTION SITE BRUISING (General disorders) | 2 | 8 | 1 | 2
INJECTION SITE SWELLING (General disorders) | 2 | 3 | 0 | 0
PYREXIA (General disorders) | 2 | 9 | 1 | 2
ADVERSE DRUG REACTIONS (General disorders) | 1 | 0 | 0 | 0
CHILLS (General disorders) | 1 | 0 | 0 | 0
ENERGY INCREASED (General disorders) | 1 | 0 | 0 | 0
FATIGUE (General disorders) | 1 | 4 | 1 | 0
INJECTION SITE ERYTHEMIA (General disorders) | 1 | 0 | 0 | 1
INJECTION SITE LACERATION (General disorders) | 1 | 0 | 0 | 0
INJECTION SITE REACTION (General disorders) | 1 | 0 | 0 | 1
INJECTION SITE ANESTHESIA (General disorders) | 0 | 0 | 0 | 1
INJECTION SITE DISCOMFORT (General disorders) | 0 | 0 | 0 | 1
INJECTION SITE IRRITATION (General disorders) | 0 | 0 | 0 | 1
INJECTION SITE MASS (General disorders) | 0 | 0 | 0 | 1
HEADACHE (Nervous system disorders) | 2 | 22 | 1 | 2
DIZZINESS (Nervous system disorders) | 1 | 7 | 2 | 1
EPILEPSY (Nervous system disorders) | 1 | 9 | 0 | 0
HYPOESTHESIA (Nervous system disorders) | 1 | 0 | 0 | 0
SOMNOLENCE (Nervous system disorders) | 1 | 8 | 2 | 3
ALTERED STATE OF CONCIOUSNESS (Nervous system disorders) | 0 | 0 | 0 | 1
POSTICTAL HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 1
CONTUSION (Injury, poisoning and procedural complications) | 1 | 9 | 1 | 0
EXCORIATION (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 0
MOUTH INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
AGITATION (Psychiatric disorders) | 2 | 4 | 1 | 0
AGGRESSION (Psychiatric disorders) | 1 | 3 | 0 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 0 | 1 | 0
CRYING (Psychiatric disorders) | 1 | 0 | 0 | 0
LOGORRHEA (Psychiatric disorders) | 1 | 0 | 0 | 0
DISORIENTATION (Psychiatric disorders) | 0 | 0 | 0 | 1
MOOD ALTERED (Psychiatric disorders) | 0 | 0 | 0 | 1
NERVOUSNESS (Psychiatric disorders) | 0 | 0 | 0 | 1
RESTLESSNESS (Psychiatric disorders) | 0 | 0 | 0 | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 | 0 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 7 | 2 | 1
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 1 | 10 | 1 | 1
MUSCLE TIGHTNESS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
YAWNING (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 1
HEART RATE INCREASED (Investigations) | 1 | 0 | 0 | 0
WEIGHT DECREASED (Investigations) | 0 | 3 | 1 | 1
INCREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 1
HYPERTENSION (Vascular disorders) | 1 | 0 | 1 | 0
FLUSHING (Vascular disorders) | 0 | 0 | 0 | 1
CONJUNCTIVAL HYPERAEMIA (Eye disorders) | 0 | 0/122 | 0 | 1
VISUAL ACUITY REDUCED (Eye disorders) | 0 | 0 | 0 | 1
EAR INFECTION (Infections and infestations) | 0 | 0 | 1 | 2
EDEMA PERIPHERAL (General disorders) | 0 | 0 | 2 | 0
ASTHENIA (General disorders) | 0 | 0 | 1 | 0
CYST (General disorders) | 0 | 0 | 1 | 0
GAIT DISTURBANCE (General disorders) | 0 | 0 | 1 | 0
PAIN (General disorders) | 0 | 0 | 1 | 0
LETHARGY (Nervous system disorders) | 0 | 5 | 0 | 0
ATAXIA (Nervous system disorders) | 0 | 3 | 1 | 0
TREMOR (Nervous system disorders) | 0 | 3 | 0 | 0
FACIAL PARESIS (Nervous system disorders) | 0 | 0 | 1 | 0
MIGRAINE (Nervous system disorders) | 0 | 0 | 1 | 0
NYSTAGMUS (Nervous system disorders) | 0 | 0 | 1 | 0
TARDIVE DYSKINESIA (Nervous system disorders) | 0 | 0 | 1 | 0
VOCAL CORD PARALYSIS (Nervous system disorders) | 0 | 0 | 1 | 0
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 | 5 | 0 | 0
THERAPEUTIC AGENT TOXICITY (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0
LACERATION (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
LIMB INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
INCISION SITE PAIN (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
JOINT INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
LIP INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
PERIORBITAL CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
INSOMNIA (Psychiatric disorders) | 0 | 3 | 3 | 0
ADJUSTMENT DISORDER (Psychiatric disorders) | 0 | 0 | 1 | 0
HALLUCINATION, VISUAL (Psychiatric disorders) | 0 | 0 | 1 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 0 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 2 | 0
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 0 | 2 | 0
COELIAC DISEASE (Gastrointestinal disorders) | 0 | 0 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 1 | 0
DIARRHEA (Gastrointestinal disorders) | 0 | 0 | 1 | 0
HEMORRHOIDS (Gastrointestinal disorders) | 0 | 0 | 1 | 0
HYPOAESTHESIA ORAL (Gastrointestinal disorders) | 0 | 0 | 1 | 0
SALIVARY GLAND MASS (Gastrointestinal disorders) | 0 | 0 | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
SCOLIOSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
WEIGHT INCREASED (Investigations) | 0 | 3 | 2 | 0
ASPIRATION TRACHEAL (Investigations) | 0 | 0 | 1 | 0
URINE OUTPUT DECREASED (Investigations) | 0 | 0 | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
HYPERLIPIDEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 1 | 0
HYPOTENSION (Vascular disorders) | 0 | 0 | 1 | 0
VISION BLURRED (Eye disorders) | 0 | 3 | 1 | 0
DIPLOPIA (Eye disorders) | 0 | 0 | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 0 | 1 | 0
SINUS TACHYCARDIA (Cardiac disorders) | 0 | 0 | 1 | 0
EAR PAIN (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 9 | 3 | 0
SINUSITIS (Infections and infestations) | 0 | 6 | 2 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 5 | 4 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 3 | 1 | 0
BRONCHITIS (Infections and infestations) | 0 | 0 | 2 | 0
INFLUENZA (Infections and infestations) | 0 | 0 | 2 | 0
OTITIS MEDIA (Infections and infestations) | 0 | 0 | 2 | 0
ACUTE SINUSITIS (Infections and infestations) | 0 | 0 | 1 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 1 | 0
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 0 | 0 | 1 | 0
SEPSIS (Infections and infestations) | 0 | 0 | 1 | 0
TONSILLITIS (Infections and infestations) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.